CLINICAL TRIAL: NCT01817114
Title: Chronic Remote Ischemic Conditioning Following Primary Percutaneous Intervention for ST-Elevated Myocardial Infarction
Brief Title: Chronic Remote Ischemic Conditioning to Modify Post-MI Remodeling
Acronym: CRIC-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University Health Network, Toronto (Other); Sunnybrook Health Sciences Centre (Other); Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000038045
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Myocardial Infarction
Keywords: Remote Ischemic Conditioning; PCI; STEMI; LAD
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Chronic Remote Ischemic Conditioning (Experimental): Remote ischemic conditioning will be induced using an AutoRIC device (occluding arm bloodflow exactly like manual bloodpressure cuff). With the participant in a supine or seated upright position, the AutoRIC device will be placed on the right arm and will inflate to a pressure of 200mmHg for 5 minutes (ischemia). The device will then auto-deflate (reperfusion), completing one cycle of ischemia-reperfusion. A total of 4 inflation and deflation cycles will occur. This will be initiated at first medical contact just prior to the performance of primary PCI in eligible subjects (RIPerC), and then repeated daily for 28 days following MI.
  Interventions: Device: Auto Remote Ischemic Conditioning (AutoRIC) device
- SHAM Remote Ischemic Conditioning (Sham Comparator): Sham conditioning will involve the AutoRIC device being placed on the right arm and will inflate to a pressure of 10mmHg for 5 minutes (ie. no limb ischemia will occur). The device will then auto-deflate, completing one cycle. A total of 4 inflation and deflation cycles will occur. This will be initiated at first medical contact just prior to the performance of primary PCI in eligible subjects (RIPerC), and then repeated daily for 28 days following MI.
  Interventions: Device: Auto Remote Ischemic Conditioning (AutoRIC) device

INTERVENTIONS:
Device: Auto Remote Ischemic Conditioning (AutoRIC) device

SUMMARY:
During a heart attack, an artery carrying blood and oxygen to the heart becomes blocked, which causes damage to the heart muscle. When possible, a clot-busting drug is given or a procedure called angioplasty is performed soon after a heart attack starts, to open up the blocked artery and restore blood flow to the heart. While this can be an effective treatment to reduce permanent damage to the heart, patients can still experience heart failure afterwards. Consequently many patients require medications to support their heart after a heart attack. Recent research has shown a new technique called Remote Ischemic conditioning or RIC, is effective at protecting the heart muscle in a heart attack. RIC is produced simply by repeated inflation and deflation of a blood pressure cuff on an arm or leg to temporarily cut off and then restore blood flow to that limb. The investigators believe this triggers the release of molecular factors that protect heart muscle. In a recent study in humans, it reduced the amount of permanent damage to the heart muscle when applied before the angioplasty procedure. The investigators recent animal studies have shown that RIC may also help the heart muscle recover after a heart attack if applied everyday during the month after a heart attack, by preventing heart failure. This is important for two reasons: first, currently the investigators can only treat heart failure with medications, and second, some people have heart attacks but are not suitable to have angioplasty and so are at greater risk of heart failure. Daily RIC may provide an easy and effective new treatment to prevent heart failure after a heart attack. This application proposes a preliminary study in humans to see if daily RIC can help heart muscle recovery after a heart attack.

ELIGIBILITY:
Inclusion Criteria:

(i) Admitted for primary PCI for STEMI involving the LAD within 12 hours of onset of symptoms. STEMI will be defined as typical ECG changes (ST segment elevation ≥2mm in 2 or more precordial leads) associated with acute chest pain or an elevation of cardiac enzymes; (ii) Antegrade TIMI 0 or 1 prior to PCI; (iii) Age ≥18 years; (iv) Informed consent from patient or next of kin.

Exclusion Criteria:

(i) Known history of diabetes; (ii) Coronary anatomy warranting emergent coronary artery bypass graft surgery; (iii) Mechanical complication of STEMI (ventricular septal rupture, free wall rupture, acute severe mitral regurgitation); (iv) Need for hemodialysis; (v) Malignancy, HIV, or central nervous system disorder; (vi) Cardiopulmonary resuscitation >15 min and compromised level of consciousness; (vii) Cardiogenic shock; (viii) Current participation in any research study involving investigational drugs or devices; (ix) Inability to safely undergo cMRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in LVEDV from baseline | 28 days post-surgery
  The primary outcome of this study will be the change from baseline in left ventricular end diastolic volume (LVEDV) at 28 days post-PCI by cardiac MRI.

SECONDARY OUTCOMES:
change in LVESV from baseline | 28 days post-surgery
  change from baseline in left ventricular end systolic volume (LVESV), ejection fraction (LVEF) and mass at 28 days post-PCI by cardiac MRI

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Redington, FRCPC, Principal Investigator — The Hospital for Sick Children; Christopher Overgaard, RCPSC, Principal Investigator — University Health Network, Toronto General Hospital
Locations (3):
- Canada (3):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario